CLINICAL TRIAL: NCT07210554
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Stapokibart Injection in Subjects With Moderate to Severe Bullous Pemphigoid
Brief Title: Study of Stapokibart Injection in Subjects With Moderate to Severe Bullous Pemphigoid
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Kangnuoxing Biopharma,Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-116201
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Bullous Pemphigoid (BP)
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: Stapokibart injection
- Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Stapokibart injection — subcutaneous injection
  Arms: Group 1
Drug: Placebo — subcutaneous injection
  Arms: Group 2

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics, and immunogenicity of Stapokibart in subjects with Moderate to Severe Bullous Pemphigoid.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study content and voluntarily sign the Informed Consent Form (ICF).
* Aged between 18 and 90 years, inclusive, regardless of gender.
* Confirmed diagnosis of bullous pemphigoid prior to randomization.
* Bullous Pemphigoid Disease Area Index (BPDAI) activity score ≥ 24 points at the screening visit and at randomization.
* Weekly average of the Pruritus Numerical Rating Scale (NRS) score ≥ 4 points at randomization.
* Karnofsky Performance Status score ≥50% at the screening visit.

Exclusion Criteria:

* Diagnosis of other forms of pemphigoid or other autoimmune blistering diseases.
* Presence of other active skin comorbidities that may interfere with the study evaluations, apart from bullous pemphigoid.
* Insufficient washout period for prior treatments.
* Any condition that, in the opinion of the investigator, would preclude the subject's participation in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-11 (Estimated); Primary Completion 2028-03-27 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving sustained complete remission (CR) at W36 | Up to 36 weeks
  Sustained complete remission (CR) defined as discontinuation of oral corticosteroid (OCS) therapy and achievement of CR on or before Week 16, no relapse during the period from OCS discontinuation up to Week 36, and no requirement for rescue therapy up to Week 36.

CONTACTS AND LOCATIONS:
Overall Officials: Hang Li, Chief physician, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China